CLINICAL TRIAL: NCT05470153
Title: The Efficacy of Continuous Positive Airway Pressure in Achieving Asthma Control in Patients With Severe Asthma and Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Siraj Omar Wali, Director of Sleep Medicine and Research Center, Professor of Medicine, King Abdulaziz University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 269-20
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Severe Asthma With Obstructive Sleep Apnea
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Asthma with Obstructive Sleep Apnea on treatment (Active Comparator): Over the following 6 months of recruiting the study population with severe asthma the following will be monitored EVERY MONTH:
  Level of asthma control: Asthma Control Test/GINA guidelines Excessive Daytime Sleepiness using Epworth Sleepiness Scale. Rate of exacerbations/hospitalization Continuous Positive Airway Pressure (CPAP) compliance: where acceptable compliance is defined as minimum of CPAP use of >/= 4 hrs/70% nights (if applicable), In one month, 3month, 6 month duration Apnea/Hypopnea Index as per CPAP reading (if applicable)
  Interventions: Device: Continuous Positive Airway Pressure
- Asthma with Obstructive Sleep Apnea whom refused treatment (No Intervention): Over the following 6 months of recruiting the study population with severe asthma the following will be monitored EVERY MONTH:
  Level of asthma control: Asthma Control Test/GINA guidelines Excessive Daytime Sleepiness using Epworth Sleepiness Scale. Rate of exacerbations/hospitalization
- Asthma without Obstructive Sleep Apnea (No Intervention): Over the following 6 months of recruiting the study population with severe asthma the following will be monitored EVERY MONTH:
  Level of asthma control: Asthma Control Test/GINA guidelines Excessive Daytime Sleepiness using Epworth Sleepiness Scale. Rate of exacerbations/hospitalization

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — For each patient with Obstructive Sleep Apnea, titration of Continuous Positive Airway Pressure (CPAP) pressure will be performed by conventional polysomnography or using auto-CPAP equipment using a validated protocol. The CPAP device should have an hour meter recording system, so that machine-on time hours could be checked at each clinical visit.
  Arms: Asthma with Obstructive Sleep Apnea on treatment

SUMMARY:
Asthma is a common heterogeneous chronic disorder of the airways, characterized by variables, usually reversible and recurring symptoms related to one or more of airflow obstruction, bronchial hyper-responsiveness, and underlying inflammation. Approximately 5-10% of asthmatics have severe or difficult to treat asthma that remains problematic despite optimal treatment. Current asthma guideline recommend investigating the presence of OSA in the cases of severe or uncontrolled asthma. Obstructive sleep apnea (OSA) is a disease that characterized by frequent narrowing or collapsed of upper airways during sleep. Recent studies have shown an overlap between Asthma and Obstructive Sleep Apnea. The mechanism of interaction between OSA and asthma is complex. Moreover, the two diseases have common comorbid conditions such as GERD and obesity which negatively impact asthma control. Polysomnography is the study of sleep using different leads, heart rate and oxygen monitor to assess the architecture of the sleep. Abnormal obstructive breathing events during monitored sleep are described according to the latest recommendation of the American Academy of Sleep Medicine. For each patient with OSA, titration of CPAP pressure will be performed by conventional polysomnography or using auto-CPAP equipment using a validated protocol. The investigators aim in this study to examine the effect of CPAP treatment in severe asthma patient with concurrent moderate and severe OSA.

DETAILED DESCRIPTION:
Asthma is a common heterogeneous chronic disorder of the airways, characterized by variables, usually reversible and recurring symptoms related to one or more of airflow obstruction, bronchial hyper-responsiveness, and underlying inflammation. the prevalence of Asthma has been increasing in the last decades, affecting over 2 million Saudis. Multiple factors had been reported in the literature that contribute to poor asthma control. Uncontrolled asthma is affecting the quality of life and is a well-known cause of mortalities. Approximately 5-10% of asthmatics have severe or difficult to treat asthma that remains problematic despite optimal treatment. It is well known that using asthma medications alone in severe asthma patients without managing the associated comorbid disease such as cardiac disease, allergic rhinitis, obesity and obstructive sleep apnea (OSA) will apprehend our goal in asthma treatment. Therefore, Current asthma guideline recommend investigating the presence of OSA in the cases of severe or uncontrolled asthma.

Obstructive sleep apnea (OSA) is a disease that characterized by frequent narrowing or collapsed of upper airways during sleep. OSA diagnoses is underestimated in the asthma population although it is considered as one of the significant comorbid disease in such populations. Overlap syndrome between Asthma and OSA has been increasing in prevalence lately, as per a recent Meta-analysis up to 50% of adults with Asthma had OSA contributing to their poor control. Yigla etal did polysomnography in a small group of patients with difficult to treat asthma who have been on long term steroid and the prevalence of OSA in this population was reported to be as high as 95%.(5) Wang et al reported that patients with asthma has a high prevalence of OSA (19.2%) compared with the control individuals (9.6%) and that OSA is associated with severe asthma exacerbation.

The mechanism of interaction between OSA and asthma is complex. Moreover, the two diseases have common comorbid conditions such as GERD and obesity which negatively impact asthma control. Using continuous positive airway pressure (CPAP) is considered to be the gold standard in the management of OSA, improving the symptoms and enhancing the quality of life. Several cohort studies of CPAP in patients with both asthma and OSA showed significant effect in achieving asthma control by improving symptoms and lung function as well as reducing the use of rescue medication. Three months of CPAP in patients with moderate to severe persistent asthma reduced serum inflammatory markers, including CRP, TNF, and IL-6. Furthermore, more recently Serrano-Pariente et al reported that asthma control, quality of life, and lung function improved after starting CPAP in asthmatics with moderate to severe OSA . However, a recent systemic review showed that CPAP therapy in asthma patient with concurrent OSA has a positive effect on quality of life and this effect is more pronounced with severe OSA in uncontrolled asthma patients.

Polysomnography (SOMNO medics plus; SOMNO medics, Randersacker, Germany) consists of continuous recordings from surface leads for electroencephalography (EEG), electrooculography, electromyography (submental and bilateral anterior tibialis muscles), electrocardiography, nasal pressure, nasal and oral airflow (thermocouple), chest and abdominal impedance belts for respiratory muscle efforts, pulse oximetry for oxygen saturation and pulse rate, a tracheal microphone for snoring and body position sensors for sleep position. PSG records are scored manually according to the American Academy of Sleep Medicine (AASM) 2012 scoring.

Abnormal obstructive breathing events during monitored sleep are described according to the latest recommendation of the AASM as a decrease in airflow by 90% or more from baseline for at least 10 seconds (apnea) and a discernible reduction in airflow of at least 30% of the pre-event baseline using nasal pressure associated with a reduction in oxygen saturation of at least 3% and/or followed by an EEG arousal (hypopnea), despite persistent chest and abdominal muscle efforts to overcome the obstruction. EEG arousal is defined according to the recommendation of the AASM. The average number of these apnea and hypopnea events per hour of sleep (i.e., the AHI) is then calculated.

Subjects with an AHI of ≥15 are categorized as having OSA, whereas those with excessive daytime sleepiness (EDS) and an AHI of ≥5 are categorized as having OSAS. Clinically diagnosed OSA (COSAS) is defined per the latest AASM recommendations (2014), i.e., A- an AHI of ≥15 determined by PSG or B- an AHI of ≥5 but <15 events, in addition to one of the following: 1) daytime sleepiness, non-restorative sleep, fatigue or insomnia symptoms; 2) incidences of waking up with gasping or choking sensations; 3) reported snoring, breathing interruptions or both during sleep; or 4) a known history of hypertension, mood or cognitive dysfunction, coronary artery disease, stroke, congestive heart failure, atrial fibrillation or diabetes mellitus. Three registered polysomnographic technologists (RPSGTs) were assigned to manually score data from these PSG studies.

For each patient with OSA, titration of CPAP pressure will be performed by conventional polysomnography or using auto-CPAP equipment using a validated protocol . The CPAP device should have an hour meter recording systems, so that machine-on time hours could be checked at each clinical visit.

Rationale The investigators aim in this study to examine the effect of CPAP treatment in severe asthma patient with concurrent moderate and severe OSA.

Study Location The study will be conducted in two tertiary hospitals in Jeddah, Saudi Arabia: King Abdulaziz Medical City and King Abdulaziz University Hospital. The patients' medical records will be reviewed to determine patients with severe asthma..

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of asthma and the classification of disease severity will be established according to the Global Initiative for Asthma (GINA) criteria. Asthma diagnosis is based either on spirometry that shows an obstructive airway defect with reversibility that has been defined as a minimum of 12% increase in the post-bronchodilator forced expiratory volume in 1 s (FEV1) and >200 mL of the FEV1, or subjects with physician-diagnosed asthma.

* Severe Asthma (defined as being on step 4 or 5 of treatment as per GINA guidelines 2019)
* All patients should not change their controller therapy for at least eight weeks before enrollment to participate in the study.
* All patients should be naïve to CPAP.

Exclusion Criteria:

* Mild or Moderate asthma according on GINA 2019
* Patients with cardiac diseases, other lung diseases (Such as COPD and restrictive lung disease), cognitive impairment that could limit the comprehension or collaboration of the subject in the study, or any severe decompensated comorbid disease
* Patients with acute asthma exacerbation within 4 weeks of recruitment
* Pregnancy
* Smoker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Determine the effect of Continuous Positive Air Pressure treatment in severe asthma patient with concurrent moderate and severe Obstructive Sleep Apnea | 6 months
  Epworth Sleepiness Scale :
  a questionnaire of 8 questions about the degree of sleepiness in different situations. Which then they grade the degree from (0)Never, (1)Slight chance, (2)Moderate chance, (3)High chance after addition of score. The results will be interpreted as follows: a score from 0-5 : considered as lower normal daytime sleepiness a score from 6-10 : considered as normal daytime sleepiness a score from 11-12 : considered as mild excessive daytime sleepiness a score from 13-15 : considered as moderate daytime sleepiness a score from 16-24 : considered as severe excessive daytime sleepiness
  The higher the score the higher chances for the patient to have excessive daytime sleepiness
Asthma Control Test (ACT) | 6 months
  contains 5 questions to assess the severity of the asthma symptoms in the last 4 weeks The results range from 5 (poor control of asthma), with a higher score 25 (complete control of asthma).
  The higher the score reflects on better control of asthma symptoms.
Asthma Symptoms Control (GINA Assessment of Asthma Control) | 6 months
  consists of 4 Yes or No questions regarding asthma symptoms in the last 4 weeks. to determine the level of asthma symptom control.
  interpretation of the result is read as:
  * Well controlled (none of the above)
  * Partly controlled (1-2 yes to the questions)
  * Uncontrolled (3-4 yes to the questions)

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Western, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No